CLINICAL TRIAL: NCT05106439
Title: Intern Health Study: 2020 Cohort Micro-Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Srijan Sen, Research Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00033029.20
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Telemedicine
MeSH Terms: interventions — Health Records, Personal

STUDY DESIGN:
Intervention Model Description: Randomization scheme
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Competition arm (Experimental): Programs with at least five interns were grouped into program-based teams. Interns within the same residency institution in programs that did not meet this criterion were grouped into institution-based teams, with a minimum of five participants per team.
  For each week, an eligible team is randomized to either competition or non-competition group with 50/50 chance. For those randomized to competition arm, teams were assigned an opponent team according to a weekly equally randomly selected rule from three options: 1. total randomization, by which the opponent team was assigned regardless of institution and specialty; 2. within-institution randomization, by which two competing teams were from the same institution; 3. within-specialty randomization, by which two paired teams were from the same specialty. For each pair of competing teams, there was a 50/50 chance that they would compete on average daily step counts or average daily sleep minutes.
  Interventions: Behavioral: Intern Health Study competition-related mobile notification; Behavioral: Intern Health Study mobile app; Behavioral: Intern Health Study mobile app competition scoreboard and history
- Non-competition group (Experimental): For each week, an eligible team is randomized to either competition or non-competition group with 50/50 chance.
  Interventions: Behavioral: Intern Health Study mobile app

INTERVENTIONS:
Behavioral: Intern Health Study competition-related mobile notification — Participants will receive three types of push notifications: 1. Alert of competition type (steps or sleep) and opponent (Sunday 9pm), 2. Competition score status update (Wednesday 9pm, Saturday 11am), and 3. Competition final results (Monday 12pm).
  Arms: Competition arm
Behavioral: Intern Health Study mobile app — The Intern Health Study mobile app is able to conduct a daily mood survey. It also aggregates and visualizes historical data on intern mood, activity, and sleep.
Behavioral: Intern Health Study mobile app competition scoreboard and history — Participant can view their current competition scoreboard and competition history at any time via the study app.
  Arms: Competition arm

SUMMARY:
The aim of this study is to evaluate the efficacy of gamified competition (delivered through a smartphone) for improving the physical activity and sleep of medical interns.

DETAILED DESCRIPTION:
Due to their high-stress workloads, medical interns tend to have lower sleep and decreased physical activity. The goal of this study is to evaluate the efficacy of gamified competition (delivered through a smartphone) for improving the physical activity and sleep of medical interns. During the study, they are teamed up by programs and institutions and competes with other teams, which aim to motivate them to have more physical activity and sleep duration during their internship year.

The primary aim of this study is to investigate whether introducing competition mechanisms into mobile health (mHealth) interventions can improve a medical intern's activity-related behavioral outcomes: daily step counts and sleep duration. The first secondary aim is to assess the time-varying competition effect on their behavioral outcomes. The second secondary aim is to evaluate how social cooperation (competing within the same institution or program) moderates the effect of competition on behavioral outcomes. The first exploratory aim is to assess the competition effect on study engagement and the second exploratory aim is to evaluate the competition effect on mental outcome, mood score.

ELIGIBILITY:
Inclusion Criteria:

* Medical intern during the 2020-2021 internship year
* Downloaded app, completed consent and filled out baseline survey prior to June 16th, 2020

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2286 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Average daily step count | 7 days
  Participants' daily step counts are recorded through a Fitbit or an apple watch. High step counts are considered a positive outcome as it indicates more physical activity.
  For teams randomized into competition arm and randomized to compete on step count, their average daily step count is compared with the average step count of the opponent team.
Average daily sleep minutes | 7 days
  Participant's nightly sleep duration (in minutes) is recorded through a Fitbit or an apple watch. High sleep duration is considered a positive outcome.
  For teams randomized into competition arm and randomized to compete on sleep duration, their average daily sleep minutes is compared with the average sleep minutes of the opponent team.

SECONDARY OUTCOMES:
Average daily mood score | 7 days
  Through the study mobile app, participants enter a mood score (scale 1-10) every day of the study. 1 corresponds to lowest mood and 10 corresponds to highest mood

CONTACTS AND LOCATIONS:
Overall Officials: Srijan Sen, M.D., Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified genomic and survey information (baseline survey, plus quarterly survey which contains the PHQ-9) will be shared with the National Institute for Mental Health (NIMH).
Supporting Information: ICF
Time Frame: Data will be made available 12 months after the end of the trial. It will be made available indefinitely after that date.
Access Criteria: The data will be shared directly with the NIMH. NIMH will apply their criteria for qualified researchers and analyses.
URL: https://www.openicpsr.org/openicpsr/project/129225/version/V1/view